CLINICAL TRIAL: NCT00822640
Title: Clinical Outcome With Attention to Functional Results One Year After Fixed or Mobile Bearing Total Knee Replacement in a Randomized Controlled Trial
Brief Title: Comparison of Rotating vs. Fixed Platform of the COLUMBUS Knee Prosthesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Dr. med. Frank Lampe, Schön Kliniken, Klinikum Eilbek
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-G-H-0301
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic; Arthrosis
Keywords: Prosthesis Design; Range of Motion, Articular; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Columbus Knee Prosthesis with rotating Platform
  Interventions: Device: Total Knee Arthroplasty
- 2 (Active Comparator): Columbus Knee Prosthesis with fixed platform
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — All patients receive the same posterior cruciate retaining implant but the tibial tray and bearing (B. Braun Aesculap Columbus CR and RP) by two experienced surgeons and will follow an identical rehabilitation regime.
  Other Names: Columbus Knee Prosthesis

SUMMARY:
A population of 100 patients randomised to rotating and fixed PE inlays in the Columbus knee prosthesis received a navigated TKR. Knee Society Score as primary endpoint, Oxford Score, and postoperative ROM after one year will be compared.

DETAILED DESCRIPTION:
Mobile bearing tibial platform designs are advocated to improve functional results of total knee replacement (TKR), and to reduce wear in the longer term. This study investigates short term functional results with two patient groups who are systematically different in the fixed or mobile tibial bearing only.

Methods: 100 knees in 97 patients are stratified according to age and gender and randomized into two groups fixed bearing (FB) with 52 knees and mobile bearing (MB) with 48 knees. All receive the same posterior cruciate retaining implant but the tibial tray and bearing (B. Braun Aesculap Columbus CR and RP) by two experienced surgeons and follow an identical rehabilitation regime. Physical examinations are performed in a double-blinded manner before the operation and three, six and twelve months thereafter, using the Oxford and Knee Society scoring systems.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective TKA
* agreement to participate in this study
* Patient age between 40 and 90 years

Exclusion Criteria:

* Malalignment of the knee to be operated of more than 20° varus or 15° valgus
* Former operations on the concerned knee (except diagnostic or therapeutic arthroscopy with only meniscus refixation or cartilage smoothing)
* Joint replacement of another joint of the same leg
* Infections in the operated joint during the follow-up period
* Thromboses during the follow-up period
* Preoperative classification according to ASA 4, 5 or 6

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 12 Months

SECONDARY OUTCOMES:
Oxford Score | 12
Range of Motion | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lampe, MD, Principal Investigator — Schön Kliniken Klinikum Eilbek
Locations (1):
- Frank Lampe, MD, Hamburg, Germany

REFERENCES:
- [Background] Buechel FF Sr, Buechel FF Jr, Pappas MJ, D'Alessio J. Twenty-year evaluation of meniscal bearing and rotating platform knee replacements. Clin Orthop Relat Res. 2001 Jul;(388):41-50. doi: 10.1097/00003086-200107000-00008. PMID 11451131
- [Background] Buechel FF Sr. Long-term followup after mobile-bearing total knee replacement. Clin Orthop Relat Res. 2002 Nov;(404):40-50. doi: 10.1097/00003086-200211000-00008. PMID 12439236
- [Background] Callaghan JJ, Squire MW, Goetz DD, Sullivan PM, Johnston RC. Cemented rotating-platform total knee replacement. A nine to twelve-year follow-up study. J Bone Joint Surg Am. 2000 May;82(5):705-11. PMID 10819281
- [Background] Callaghan JJ. Mobile-bearing knee replacement: clinical results: a review of the literature. Clin Orthop Relat Res. 2001 Nov;(392):221-5. doi: 10.1097/00003086-200111000-00027. PMID 11716386
- [Background] Callaghan JJ, Insall JN, Greenwald AS, Dennis DA, Komistek RD, Murray DW, Bourne RB, Rorabeck CH, Dorr LD. Mobile-bearing knee replacement: concepts and results. Instr Course Lect. 2001;50:431-49. PMID 11372345
- [Background] Catani F, Benedetti MG, De Felice R, Buzzi R, Giannini S, Aglietti P. Mobile and fixed bearing total knee prosthesis functional comparison during stair climbing. Clin Biomech (Bristol). 2003 Jun;18(5):410-8. doi: 10.1016/s0268-0033(03)00044-5. PMID 12763437
- [Background] Chiu KY, Ng TP, Tang WM, Lam P. Bilateral total knee arthroplasty: One mobile-bearing and one fixed-bearing. J Orthop Surg (Hong Kong). 2001 Jun;9(1):45-50. doi: 10.1177/230949900100900109. PMID 12468843
- [Background] Emerson RH Jr, Hansborough T, Reitman RD, Rosenfeldt W, Higgins LL. Comparison of a mobile with a fixed-bearing unicompartmental knee implant. Clin Orthop Relat Res. 2002 Nov;(404):62-70. doi: 10.1097/00003086-200211000-00011. PMID 12439239
- [Background] Grodzki T, Haak H, Behrendt R, Merk H, Krauspe R. [Prospective randomized comparative study of early functional outcome of 2 knee joint endoprosthesis systems--rotation plateau versus fixed polyethylene inlay]. Z Orthop Ihre Grenzgeb. 2001 Sep-Oct;139(5):393-6. doi: 10.1055/s-2001-17980. German. PMID 11605289
- [Background] Kim YH, Kook HK, Kim JS. Comparison of fixed-bearing and mobile-bearing total knee arthroplasties. Clin Orthop Relat Res. 2001 Nov;(392):101-15. doi: 10.1097/00003086-200111000-00013. PMID 11716371
- [Background] Price AJ, Rees JL, Beard D, Juszczak E, Carter S, White S, de Steiger R, Dodd CA, Gibbons M, McLardy-Smith P, Goodfellow JW, Murray DW. A mobile-bearing total knee prosthesis compared with a fixed-bearing prosthesis. A multicentre single-blind randomised controlled trial. J Bone Joint Surg Br. 2003 Jan;85(1):62-7. doi: 10.1302/0301-620x.85b1.13233. PMID 12585579
- [Background] Vertullo CJ, Easley ME, Scott WN, Insall JN. Mobile bearings in primary knee arthroplasty. J Am Acad Orthop Surg. 2001 Nov-Dec;9(6):355-64. doi: 10.5435/00124635-200111000-00001. PMID 11730328
- [Derived] Marques CJ, Daniel S, Sufi-Siavach A, Lampe F. No differences in clinical outcomes between fixed- and mobile-bearing computer-assisted total knee arthroplasties and no correlations between navigation data and clinical scores. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1660-8. doi: 10.1007/s00167-014-3127-x. Epub 2014 Jun 15. PMID 24929659